CLINICAL TRIAL: NCT06969794
Title: Single-center, Single Group, Randomized, Superiority Pivotal Clinical Study to Evaluate the Efficacy and Safety of Artificial Intelligence-based Upper Gastrointestinal Endoscopy Image Diagnosis Aid Software
Brief Title: Single-center, Randomized, Superiority Pivotal Clinical Study to Evaluate the Efficacy of Artificial Intelligence-based Upper Gastrointestinal Endoscopy Image
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, PI, Chuncheon Sacred Heart Hospital
Other Study IDs: AI RCT2
Record Dates: First submitted 2025-04-25; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gastric Neoplasm; Gastric Lesion; Artificial Intelligence
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will conduct a single-center retrospective study at a university hospital. A total of 3,385 gastroscopic white-light images from patients with pathologically confirmed findings will be analyzed. The AI software will automatically identify images as non-neoplastic or neoplastic (low-grade dysplasia, high-grade dysplasia, early gastric cancer with mucosal or submucosal invasion, or advanced gastric cancer) and highlighted lesion locations. Two experienced endoscopists will independently review the same image set without AI assistance for comparison. Primary outcomes are sensitivity and specificity of the AI in detecting gastric neoplasms (by category and overall), and the localization accuracy measured by the localization receiver operating characteristic (LROC) curve area. Secondary outcomes is includes comparison of the AI's diagnostic performance with that of endoscopists.

DETAILED DESCRIPTION:
We will conduct a single-center retrospective study at a university hospital. A total of 3,385 gastroscopic white-light images from patients with pathologically confirmed findings will be analyzed. The AI software will automatically identify images as non-neoplastic or neoplastic (low-grade dysplasia, high-grade dysplasia, early gastric cancer with mucosal or submucosal invasion, or advanced gastric cancer) and highlighted lesion locations. Two experienced endoscopists will independently review the same image set without AI assistance for comparison. Primary outcomes are sensitivity and specificity of the AI in detecting gastric neoplasms (by category and overall), and the localization accuracy measured by the localization receiver operating characteristic (LROC) curve area. Secondary outcomes is includes comparison of the AI's diagnostic performance with that of endoscopists.

Inclusion criteria:

Age 19 or older At least one gastric lesion biopsied with a definitive pathological diagnosis Availability of high-quality white-light endoscopy images of the lesion and surrounding mucosa

Exclusion criteria:

Poor-quality images (e.g., out of focus or obscured) Lack of histopathological confirmation of the lesion

Each image will be paired with a reference standard diagnosis based on the pathology result for that lesion or region.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 or older
* At least one gastric lesion biopsied with a definitive pathological diagnosis
* Availability of high-quality white-light endoscopy images of the lesion and surrounding mucosa

Exclusion Criteria:

* Poor-quality images (e.g., out of focus or obscured)
* Lack of histopathological confirmation of the lesion

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 3,385 endoscopic images were collected from patients who underwent gastroscopy at our institution (Chuncheon Sacred Heart Hospital from 2010 to 2017) and had adequate reference standards. Images were selected to include both neoplastic lesions and non-neoplastic findings. Inclusion criteria were images of gastric lesions that had definitive histopathology diagnoses (from endoscopic biopsy or resection) of one of five severity categories: LGD, HGD, EGC-M (mucosal early gastric carcinoma), EGC-SM (submucosal invasive early carcinoma), or AGC (advanced gastric cancer). Additionally, a set of non-neoplastic images (normal or benign findings with negative biopsies) was included as controls.
Sampling Method: Non-Probability Sample
Enrollment: 3385 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
AI performance | Day 1
  sensitivity and specificity of the AI in detecting gastric neoplasms (by category and overall), and the localization accuracy measured by the localization receiver operating characteristic (LROC) curve area.

SECONDARY OUTCOMES:
comparison of the AI's diagnostic performance with that of endoscopists. | Day 1
  Secondary outcomes included comparison of the AI's diagnostic performance with that of endoscopists. (sensitivity and specificity of the AI in detecting gastric neoplasms (by category and overall), and the localization accuracy measured by the localization receiver operating characteristic (LROC) curve area.)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, MD, PhD, Principal Investigator — HALLYM UNIVERSITY COLLEGE OF MEDICINE, Korea
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, Gangwon-do, South Korea